CLINICAL TRIAL: NCT04884906
Title: A Single-arm, Single-center, Open, Prospective Phase II Clinical Study of Camrelizumab Combined With Radiotherapy and Chemotherapy for the Treatment of Recurrent or Metastatic Cervical Cancer
Brief Title: Camrelizumab Combined With Radiotherapy and Chemotherapy for the Treatment of Recurrent or Metastatic Cervical Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: E20210044
Record Dates: First submitted 2021-05-11; First posted 2021-05-13 (Actual); Last update posted 2021-05-13 (Actual); Status verified 2021-05

CONDITIONS: Locally Advanced Cervical Cancer
MeSH Terms: interventions — camrelizumab; Radiotherapy; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Camrelizumab combined with radiotherapy and chemotherapy (Experimental)
  Interventions: Biological: Camrelizumab; Radiation: radiotherapy; Drug: Albumin Paclitaxel; Drug: Cisplatin

INTERVENTIONS:
Biological: Camrelizumab — 200mg/m2, iv, d1, Q3W, a total of 6 cycles
Radiation: radiotherapy — 1.8-2.15Gy/time (radiotherapy started on the 8th day of camrelizumab treatment), a total of 28 times (5 times a week), a total of 50.4-60.2Gy.
Drug: Albumin Paclitaxel — 260mg/m2, iv, d1, Q3W, a total of 6 cycles
Drug: Cisplatin — 80-120mg/m2, iv, d1-3, Q3W, a total of 6 cycles

SUMMARY:
To evaluate the effectiveness and safety of camrelizumab combined with radiotherapy and chemotherapy for recurrent or metastatic cervical cancer

DETAILED DESCRIPTION:
This study is a single-arm, single-center, open, prospective phase II clinical study, the main purpose of which is to evaluate the effectiveness and safety of camrelizumab combined with radiotherapy and chemotherapy for recurrent or metastatic cervical cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years old and ≤75 years old;
2. ECOG score 0-1 level;
3. Cervical cancer diagnosed pathologically, cervical cancer that has recurred or metastasized after at least first-line chemotherapy or surgery;
4. Genetic testing: PD-L1≥1%;
5. The expected survival period is ≥6 months;
6. The functional level of major organs must meet the following requirements:

   Blood routine: ANC≥1.5×109/L; PLT≥90×109/L; Hb≥90 g/L; Blood biochemistry: TBIL≤2.5×ULN; ALT and AST≤1.5×ULN; BUN and Cr ≤1.5×ULN;
7. Heart color Doppler ultrasound: LVEF≥50%;
8. 12-lead electrocardiogram: QT interval (QTcF) corrected by Fridericia method <450 ms for males and <470 ms for females;
9. No blood transfusion within 2 weeks before screening;
10. For female subjects who have not undergone menopause or have not undergone surgical sterilization, during the treatment period and at least 7 months after the last administration in the study treatment, agree to abstain from sex or use an effective method of contraception;
11. Volunteer to join the study, sign informed consent, have good compliance and are willing to cooperate with follow-up.

Exclusion Criteria:

1. Have received previous anti-tumor therapy or radiotherapy for any malignant tumor, excluding cured cervical carcinoma in situ, basal cell carcinoma or squamous cell carcinoma and other malignant tumors;
2. Previously received camrelizumab or other PD-1/PD-L1 treatments and cannot be included in the group; the subject is known to have been exposed to macromolecular protein preparations, or is known to be against any carrelizumab, or Subjects are allergic to the chemotherapeutic ingredients used during neoadjuvant treatment;
3. At the same time receive anti-tumor therapy in other clinical trials, including endocrine therapy, bisphosphonate therapy or immunotherapy;
4. In the 4 weeks before randomization, have received major surgical operations not related to cervical cancer, or the subject has not fully recovered from such surgical operations.
5. Those who are known to have a history of allergies to the drug components of this program;
6. A history of immunodeficiency, including a positive HIV test, or other acquired or congenital immunodeficiency diseases, or a history of organ transplantation.
7. Have ever suffered from any heart disease, including: (1) angina pectoris; (2) arrhythmia requiring medical treatment or clinical significance; (3) myocardial infarction; (4) heart failure; (5) any investigator Other heart diseases judged to be unsuitable for participating in this test.
8. Female patients during pregnancy and lactation, female patients with fertility and a positive baseline pregnancy test, or female patients of childbearing age who are unwilling to take effective contraceptive measures during the entire trial period.
9. According to the judgment of the investigator, there are concomitant diseases (including but not limited to high blood pressure, severe diabetes, active infection, thyroid disease, etc.) that seriously endanger the safety of the patient or affect the completion of the study;
10. Inability to swallow, chronic diarrhea and intestinal obstruction, there are many factors that affect the administration and absorption of drugs.
11. The researcher believes that the subject is not suitable for participating in any other situations in this research.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2020-11-01 (Actual); Primary Completion 2022-11-01 (Estimated); Study Completion 2024-11-01 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) | 2 year
  The objective remission rate refers to the proportion of patients whose tumors have shrunk to a certain amount and maintained for a certain period of time, including cases of complete remission and partial remission

SECONDARY OUTCOMES:
Progression-free survival（PFS） | 2 year
  The period of time between when a patient with neoplastic disease receives treatment and when the disease progresses or death from any cause occurs
Overall survival（OS） | 2 year
  The time from the patient's confirmation of the disease to death due to any cause
Disease control rate（DCR） | 2 year
  Refers to the proportion of patients whose tumors have shrunk or stabilized for a certain period of time, including complete remission (CR), partial remission (PR) and stable (SD) cases
Adverse reaction rate | 2 year
  Harmful and unrelated reactions that occur when normal doses of drugs are used to prevent, diagnose, treat diseases or regulate physiological functions
Patient quality of life | 2 year
  Comprehensively evaluate the pros and cons of life by filling in the questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- TianjinCIH, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: No